CLINICAL TRIAL: NCT07371806
Title: THE EFFECT OF A MINDFULNESS-BASED STRESS REDUCTION PROGRAM ON QUALITY OF LIFE , ANXIETY AND EMPOWERMENT LEVELS IN WOMEN WITH CORONARY ARTERY DISEASE
Brief Title: EFFETCS OF MİNDFULNESS-BASED STRESS REDUCTION İN WOMEN WİTH CORONARY ARTERY DİSEASE
Acronym: MBSR-CADWOMEN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Collaborators: Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, HATİCE PENEKLİ, HATİCE PENEKLİ, PhD Candidate, Faculty of Nursing, Institute of Health Sciences, Erciyes University, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ErciyesU-SBF-HP-01
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: Coronary artery disease; Mindfulness-based intervention; Quality of life
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: The study includes one intervention group and one control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Intervention Group (Experimental): Participants in the intervention group will take part in an 8-week mindfulness-based program designed to cultivate awareness related to anxiety, psychological resilience, and quality of life in women with coronary artery disease.
  Interventions: Behavioral: Mindfulness-Based Intervention Program
- Standard Care in Women with Coronary Artery Disease (No Intervention): Participants in the control group will receive standard care, including routine medical follow-up and discharge education, without any structured intervention.

INTERVENTIONS:
Behavioral: Mindfulness-Based Intervention Program — This intervention is an 8-week structured mindfulness-based program designed to cultivate awareness related to anxiety, psychological resilience, and quality of life in women with coronary artery disease. The program includes meditation, breathing, and mindfulness exercises, distinguishing it from the standard care received by the control group.
  Arms: Mindfulness-Based Intervention Group

SUMMARY:
Coronary artery disease (CAD) is a common cardiovascular condition characterized by the narrowing or blockage of the coronary arteries that supply oxygen-rich blood to the heart muscle. CAD represents a significant cause of morbidity and mortality, particularly among individuals aged 40 and older, affecting millions of men and women worldwide. Patients with CAD experience not only physical symptoms but also psychological challenges, including stress and anxiety, which can negatively impact quality of life. In recent years, mindfulness-based interventions have emerged as scientifically supported approaches to help individuals with chronic diseases manage stress and enhance emotional regulation skills. While the existing literature includes studies evaluating the effects of mindfulness-based interventions in CAD and other cardiovascular conditions, most investigations address mixed patient populations and do not thoroughly examine sex-specific differences. Notably, women with CAD may experience symptoms and psychological effects differently than men. Therefore, there is a need for tailored, comprehensive intervention models that address the multidimensional needs of female patients, including stress management, anxiety reduction, and empowerment. This study aims to evaluate the effectiveness of mindfulness-based interventions in women with CAD, providing a targeted approach that addresses both clinical and psychosocial outcomes. The findings are expected to offer valuable insights into improving quality of life and enhancing coping strategies for women living with chronic cardiovascular disease.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is a prevalent cardiovascular condition that develops as a result of narrowing or blockage of the coronary arteries supplying blood to the heart, significantly affecting the cardiovascular system. CAD is recognized as a major cause of morbidity and mortality, particularly among individuals aged 40 and older. According to 2024 data from the British Heart Foundation (BHF), approximately 110 million men and 80 million women worldwide are affected by CAD, with the disease accounting for one in every six deaths globally. Similarly, data from the Turkish Statistical Institute, indicate that circulatory system diseases represent 36% of total deaths in Turkey, with 42.9% of these deaths attributable to ischemic heart diseases. CAD not only adversely impacts individual health but also imposes a significant burden on public health and healthcare systems. Its high prevalence, associated morbidity and mortality, long-term and costly treatment requirements, and the resulting decline in quality of life position CAD as a critical public health priority. Affecting millions of men and women worldwide, CAD leads not only to physical symptoms but also to psychological challenges that reduce quality of life. Stress, anxiety, and depressive symptoms are common psychosocial issues among patients with CAD and can complicate the management of chronic disease. In managing chronic illnesses, it is essential to enhance individuals' stress-coping skills, improve emotional regulation, and strengthen psychological resilience. In recent years, mindfulness-based interventions have emerged as scientifically supported approaches to achieve these objectives. Mindfulness and other awareness-based programs have been shown to help individuals cope with stress, manage anxiety, and improve psychological resilience. Existing literature includes studies evaluating the effects of mindfulness-based interventions in CAD and other cardiovascular conditions. However, most of these studies examine mixed patient populations and do not thoroughly investigate sex-specific differences. Notably, women with CAD experience symptoms, psychological stress, and quality-of-life challenges differently than men. Therefore, there is a clear need for tailored, targeted intervention models specifically designed for female patients with CAD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with coronary artery disease (CAD) for at least 1 month.
* Score of 14 or higher on the Short Form of the State-Trait Anxiety Inventory (STAI-SF) at baseline.
* At least primary school education.
* Age between 18 and 50 years.
* Sexually active.
* Having an active social network.

Exclusion Criteria:

* Individuals with hearing or language impairments that would hinder communication.
* Women who have entered menopause.
* Women with psychiatric disorders.

Discontinuation Criteria:

* Participants who choose to withdraw from the study.
* Participants who miss two intervention sessions.
* Participants with incomplete data on study forms.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only female patients with coronary artery disease are eligible to participate in the study.
Enrollment: 70 (Estimated)
Dates: Start 2026-04-15 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Cardiac Quality of Life Scale | Baseline and at the end of the 8-week program
  The Heart Quality of Life Scale (HeartQoL) is a reliable instrument developed to assess quality of life in individuals with ischemic heart disease (Oldridge, 2014). The scale consists of 14 items, with 10 assessing physical aspects and 4 assessing emotional aspects. Each item is scored from 0 to 3, with higher scores indicating better quality of life. It can be applied to individuals aged 18 and above. Turkish validity and reliability were established by Duğan (2018).

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory - Short Form (STAI-SF) | Baseline and at the end of the 8-week program
  The State-Trait Anxiety Inventory - Short Form (STAI-SF) is a reliable tool developed to assess general anxiety levels in individuals (Spielberger et al., 1970). Its Turkish adaptation was made by Öner and Le Compte (1985). The short form was later developed by Zsido et al. (2020) and consists of 5 items using a 4-point Likert scale. Scores of 14 or higher indicate clinically significant anxiety. The internal consistency ranges between 0.83-0.86, and its Turkish validity and reliability have been established (Döner et al., 2021). The scale can be applied to individuals aged 18 and above.

OTHER OUTCOMES:
Coronary Artery Disease Empowerment Scale | Baseline and at the end of the 8-week program
  The Coronary Artery Disease Empowerment Scale (CADES) is a reliable tool developed to assess patients' ability to manage their health and their empowerment levels (Kim et al., 2021). The scale consists of 24 items across three subscales: Autonomy (12 items), Emotional Self-Control (6 items), and Perceived Personal Competence in Disease Management (6 items). Items are rated on a 5-point Likert scale; higher scores indicate greater empowerment. Turkish validity and reliability were established by Çetin and Arslan (2023). The scale can be applied to individuals aged 18 and above.

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri Şehir Hastanesi, Kayseri, Türki̇ye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant information will not be shared at this time, as the study has not yet started and confidentiality must be maintained.